CLINICAL TRIAL: NCT04695340
Title: Effect of Psyllium (Plantago Ovata) on Digestive Disorders in Familial Amyloidosis
Acronym: Psyllium
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No inclusion during the authorised period, no extension is possible again
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-PP-12
Record Dates: First submitted 2021-01-04; First posted 2021-01-05 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Familial Amyloidosis
MeSH Terms: conditions — Amyloidosis, Familial | interventions — Psyllium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Familial amyloidosis patients (Experimental): Familial amyloidosis patients with gastro-intestinal pain receiving Psyllium
  Interventions: Dietary Supplement: Psyllium

INTERVENTIONS:
Dietary Supplement: Psyllium — Psyllium is given to patients

SUMMARY:
Familial amyloidosis is a rare disease that mainly affects the nerves and heart, but also more rarely the eyes and kidneys. This disease is due to a mutation in the gene encoding the synthesis of transthyretin, resulting in a modification of the translated protein. This abnormal protein and its derivatives are deposited in the form of a toxic "amyloid" substance in tissues and organs, altering their functions, particularly in the gastrointestinal tract.

From a gastrointestinal perspective, different treatments can be proposed in the absence of specific recommendations for familial amyloidosis. The hygienic and dietary measures consist of avoiding tobacco, alcohol and carbonated drinks, limiting fatty meals rich in poorly digestible fibers, and splitting meals. If this fails, metoclopramide and domperidone are suggested. As a second-line erythromycin, can be used with caution because of cardiac risks and drug interactions. Polyethylene glycol-based osmotic laxatives can be used to treat constipation. Alternating diarrhea and constipation can be treated with ispaghul-based laxatives, aiming at transit regulation. Finally, refractory diarrhea can be treated with the administration of loperamide. If this fails, treatment with a somatostatin analogue may be offered.

However, all these treatments can present significant side effects, therefore natural alternatives are often sought. Psyllium in particular regulates transit by normalizing stool consistency: it is effective against digestive disorders such as constipation, but it is also effective in the event of diarrhea. It allows the formation of a viscous gel by the hydrophilicity of polysaccharides macromolecules, increasing the fecal bowl which stimulates peristalsis and facilitates defecation. The WHO has recognized that Psyllium is superior to wheat bran in the treatment of irritable bowel syndrome.

The main objective of the study is to assess the effect of daily Psyllium administration on digestive quality of life in familial amyloidosis patients who suffer from digestive disorders.

ELIGIBILITY:
Inclusion criteria:

* male or female age ≥ 18
* suffering from familial amyloidosis confirmed by: i) the presence of a specific mutation in transthytetin gene and/or ii) amyloid deposits immunostained for transthyretin in a tissue biopsy
* stage 1 or 2 on the familial amyloid polyneuropathy scale
* receiving a stable dose for at least 3 months if treated with Patisaran® and inotersen (Tegsedi®),
* suffering from gastro intestinal pain ≥ 4 on Visual Analog Scoale (VSA)
* affiliated to social security
* able to understand the inform consent form
* if women of child bearing age, using an effective birth control method for the period of study participation

Exclusion criteria:

* allergic to Psyllium
* intestinal or esophageal stenosis or any other type of real or suspected gastrointestinal obstruction
* protection by law under guardianship, or who cannot participate in a clinical study under Article L. 1121-16 of the French Code of Public Health
* participation in the last 3 months in a clinical research study in which he / she has been exposed to a pharmaceutical product or a medical device
* treatment with tafamidis (Vyndaqel®)
* concomitant intake of food supplements containing zinc, iron, calcium, magnesium or vitamin B12,
* contraindication to taking Psyllium, e.g. fecal impaction, gastrointestinal obstruction, esophageal or intestinal stenosis or dysphagia to liquids
* stage 0 or 3 on the familial amyloid polyneuropathy scale
* pregnant or breastfeeding female patient (a urine pregnancy test will be performed for women of childbearing age)
* any pathology or concomitant treatment that may interfere with the progress of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Effect of Psyllium administration on digestive quality of life in familial amyloidosis patients | 6 months
  The effect of Psyllium administration on digestive quality of life in familial amyloidosis patients will be evaluated at 6 months using the Gastrointestinal Quality of Life index (GIQLI)

SECONDARY OUTCOMES:
Effect of Psyllium administration on global quality of life in familial amyloidosis patients | 6 months
  The effect of Psyllium administration on global quality of life in familial amyloidosis patients will be evaluated at 6 months using the Norfolk Quality of Life - questionnaire
Effect of Psyllium administration on motor function in familial amyloidosis patients | 6 months
  The effect of Psyllium administration on motor function in familial amyloidosis patients will be evaluated at 6 months using the Neuropathy Impairment Score Lower Limb tests (0 to 88; 0 is defined as a normal status)
Effect of Psyllium administration on gastro intestinal pain in familial amyloidosis patients | 6 months
  The effect of Psyllium administration on gastro intestinal pain in familial amyloidosis patients will be evaluated at 6 months using the visual analogy scale (0 to 10; 0 is defined as no pain status)
Effect of Psyllium administration on stool density in familial amyloidosis patients | 6 months
  The effect of Psyllium administration on stool density in familial amyloidosis patients will be evaluated at 6 months using the Bristol score (1 to 7; 1-2 is defined as a constipation status, 3-4 is the most regular status, 5-7 is defined by diarrheas)
Adverse effects of Psyllium administration in familial amyloidosis patients | 6 months
  Adverse effects of Psyllium administration in familial amyloidosis patients will be recorded thoughout the study

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Nice, Nice, Provence-Alpes-Côte d'Azur Region, France

IPD SHARING:
Plan to Share IPD: No